CLINICAL TRIAL: NCT06541990
Title: HARMONY: A Psychoeducational Intervention to Reduce Psychological Distress and Improve Quality of Life for Patients With Hepatocellular Carcinoma
Brief Title: Psychoeducational Intervention for Patients With Hepatocellular Carcinoma
Acronym: HARMONY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kelsey S. Lau-Min, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-371
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Harmony Hard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HARMONY (Experimental): HARMONY is a psychoeducational intervention that consists of three one-on-one coaching sessions and a structured session workbook.
  Interventions: Behavioral: HARMONY
- Enhanced usual care (Active Comparator): The enhanced usual care condition consists of a curated list of supportive care services for patients with HCC.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: HARMONY — A psychoeducational intervention for patients with HCC
  Arms: HARMONY
Other: Enhanced usual care — A supportive care resource guide
  Arms: Enhanced usual care

SUMMARY:
This study aims to refine and pilot test HARMONY, a psychoeducational intervention for patients with newly diagnosed hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
There are two parts of this study. Study Part 1 is an open pilot study to refine HARMONY prior to larger-scale testing in a randomized controlled trial (RCT) setting. Study Part 1 is purely descriptive, as the investigators will use the data to refine HARMONY before proceeding to Study Part 2.

Study Part 2 is a pilot RCT to assess the feasibility and acceptability of conducting a randomized trial of HARMONY versus enhanced usual care. Participants will complete a baseline survey and then be randomized to HARMONY versus enhanced usual care (a supportive care resource guide). This record reflects the clinical trial component (Study Part 2), as feasibility and acceptability outcomes will be collected for this phase only.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* New diagnosis of HCC within the last six months
* Ability to complete study procedures English

Exclusion Criteria:

* Incidentally diagnosed with HCC after liver transplantation
* Significant uncontrolled hepatic encephalopathy, cognitive impairment, or psychiatric disorder which will interfere with study participation
* Patients near the end of life for whom hospice is recommended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: study enrollment rate | 10 weeks
  ≥40% enrollment among consecutive eligible patients

SECONDARY OUTCOMES:
Feasibility: intervention completion rate | 10 weeks
  ≥50% completion of 2/3 intervention sessions in the HARMONY arm
Acceptability | 10 weeks
  ≥70% of patients in the HARMONY arm reporting Client Satisfaction Questionnaire-8 (CSQ-8) scores at or above the midpoint score of 20 on a scale from 8-32

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No